CLINICAL TRIAL: NCT05235204
Title: Early Foley Catheter Removal After Diverticular Colovesical Fistula Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karim Alavi (Other)
Responsible Party: Sponsor-Investigator, Karim Alavi, Associate Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00016345
Record Dates: First submitted 2021-12-16; First posted 2022-02-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Colovesical Fistula
MeSH Terms: conditions — Intestinal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foley catheter removal day 2 or 3 post-operative procedure (Experimental): According to review of internal clinical practices, the average duration of catheterization after Colovesical Fistula (CVF) repair is 10.8 days after CVF repair. The intervention in this study removes the Foley Catheter at 2 to 3 days post CVF repair.
  Interventions: Procedure: Removal of Foley Catheter 2 to 3 days post Colovesical Fistula (CVF) repair surgery

INTERVENTIONS:
Procedure: Removal of Foley Catheter 2 to 3 days post Colovesical Fistula (CVF) repair surgery — According to review of internal clinical practices, the average duration of catheterization after Colovesical Fistula (CVF) repair is 10.8 days after CVF repair. The intervention in this study removes the Foley Catheter at 2 to 3 days post CVF repair.

SUMMARY:
Patients undergoing surgical repair of colovesical fistula will have have "early" (post-operative day 3) cystogram and removal of bladder catheter. Outcomes from the "early" group will be compared to historical "late" group data to determine if early bladder catheter removal is safe.

DETAILED DESCRIPTION:
There is defined time for foley/bladder catheter removal after colovesical fistula repair in the current surgical literature. This study will be a prospective cohort study evaluating outcomes after early foley catheter removal (on post-operative day 3), specifically bladder leak, 30-day readmissions and adverse events. This cohort will be compared to a retrospective "late" group, who had foley catheter removal later in their hospital course.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Undergoing surgical repair of diverticular colovesical fistula

Exclusion Criteria:

* Patients with active and untreated genitourinary cancers
* Subjects with known or suspected Inflammatory Bowel Disease as the cause of colovesical fistula.
* Individuals who are not expected to regain normal bladder function after surgery as defined by either pre-existing bladder dysfunction with chronic indwelling urinary catheter, supra-pubic catheter, or surgical urinary diversion
* Individuals who require re-operation prior to Foley removal
* Adults unable to consent
* Pregnant women
* Prisoners
* Individuals who are not yet adults (infants, children, teenagers less than 18 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Presence of positive urine leak on post-operative day 3 cystogram | up to 3 days post surgery
  Participants cystograms will be reviewed to detect positive urine leak, 2 to 3 days post surgery.

SECONDARY OUTCOMES:
Foley catheter re-insertion | up to 5 days post-surgery
  Participants who will require re-insertion of the foley catheter once it is removed on post-operative day 3
Re-operations within 30 days of initial surgery | up to 30 days post discharge
  Patients who have required return to the OR within 30 days after discharge.
Hospital re-admission | up to 30 days post- discharge
  Patients who have required readmission to the hospital within 30 days after discharge.
Symptomatic post-operative urinary tract infection | up to days post discharge
  Patients who have had a symptomatic urinary tract infection within 30 days after discharge.
Post operative urinary sepsis | up to 30 days post discharge
  Patients who have urinary sepsis either prior to discharge or within 30 days after discharge.
Recurrence of colovesical fistula | up to 30 days post-discharge
  Patients who had recurrence of their colovesical fistula within 30 days of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: KArin Alavi, MD, MPH, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Memorial Medical Center Memorial Campus, Worcester, Massachusetts, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT05235204/ICF_000.pdf